CLINICAL TRIAL: NCT01698138
Title: Prevention of Bladder Dysfunction in Acute Spinal Cord Injury. A Double-blind, Randomized, Placebo-controlled Study to Explore the Effect of Early Treatment With Onabotulinumtoxin A on Development of Detrusor Overactivity
Brief Title: Prevention of Bladder Dysfunction in Acute Spinal Cord Injury
Acronym: BOT-SCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Sunnaas Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Lars Frich, MD, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012/1151
Record Dates: First submitted 2012-09-26; First posted 2012-10-02 (Estimated); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Spinal Cord Injuries; Urinary Bladder, Overactive
Keywords: Spinal cord injury; Neurogenic overactive bladder; Onabotulinum toxin A; Prevention; Botulinum Toxins, Type A
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 30 transurethral injections, each of 1 ml solution containing NaCl.
  Interventions: Drug: Placebo
- Onabotulinumtoxin A (Active Comparator): 30 transurethral injections, each of 1 ml solution containing 300 U Onabotulinumtoxin A (Botox ®, "Allergan") in 30 ml of NaCl 0.9 %.
  Interventions: Drug: Onabotulinumtoxin A

INTERVENTIONS:
Drug: Onabotulinumtoxin A — 30 transurethral injections, each of 1 ml solution containing 300 U Onabotulinumtoxin A (Botox ®, "Allergan") in 30 ml of NaCl 0.9 %.
  Other Names: Botox ®, "Allergan"
  Arms: Onabotulinumtoxin A
Drug: Placebo — 30 transurethral injections, each of 1 ml solution containing NaCl.
  Other Names: NaCl
  Arms: Placebo

SUMMARY:
This study is a double blind, randomized, placebo controlled trial to explore the effect of early treatment with Onabotulinumtoxin A in patients with acute complete motor spinal cord injury (SCI) on the development of neurogenic detrusor overactivity (NDO). A total of 20 patients will be randomized to intra-detrusor injection of 300 U Onabotulinumtoxin A in 30 ml NaCl 0.9 % or placebo with 30 ml NaCl 0.9 %. Bladder biopsies will be obtained in the same procedure. The treatment will be repeated after three months. All included patients will be evaluated with urodynamic examinations. Follow-up is 12 months after the first treatment. The primary endpoint of the study is development of NDO.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented acute, motor complete C6 to Th11 spinal cord injury
* Patients can be included in the study less than four weeks after injury
* Male or female, aged 18 to 80 years old
* Patient weight > 40 kg
* Patient is able and willing to sign informed consent
* Patient is able to complete all study requirements

Exclusion Criteria:

* Neurogenic detrusor overactivity with contractions greater than 40 cm H2O at first visit
* History or evidence of previous urological abnormalities, disease or surgery, except bladder dysfunction after spinal cord injury
* History of haematuria or ongoing haematuria, if the hematuria is determined to be a pathologic condition or is uninvestigated
* Pregnancy or females of childbearing potential unwilling to use a reliable form of contraception
* Breastfeeding
* Known allergy to Onabotulinumtoxin A
* Grave psychiatric disorder
* Use of anti-platelet or anti-coagulant other than low molecular weight heparin (LMWH) or acetylsalicylic acid
* Haemophilia or other clotting disorders that cause bleeding diathesis
* Treatment with antimuscarinic medication within 3 months of randomization
* Treatment with botulinum toxin of any serotype within 3 months of randomization
* Patient has been immunized for any botulinum toxin serotype
* Patient has any medical condition that may put the patient at increased risk with exposure to botulinum toxin including diagnosed myasthenia gravis, Eaton-Lambert syndrome or amyotrophic lateral sclerosis
* Patient has any condition or situation, which, in the investigator's opinion, puts the patient at significant risk, could confound the study results, or may interfere significantly with the patient's participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-09; Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Presence of neurogenic detrusor overactivity during cystometry, defined as contractions with amplitudes above 40 cm H2O. | 12 months

SECONDARY OUTCOMES:
Urodynamic parameters | 12 months
  Maximal detrusor pressure (cmH2O), maximal bladder capacity (ml), compliance (ΔcmH2O/Δml), and occurrence of DSD.
Quality of life (QOL) in the treated group compared to the placebo group 12 months after first treatment. | 12 months
Occurrence of complications. | 12 months

OTHER OUTCOMES:
Detrusor pathophysiology | 12 months
  Differences in levels of transmitters and receptors relevant to development of bladder dysfunction, measured in urine samples and bladder biopsies, to gain knowledge of the pathophysiology behind neurogenic detrusor overactivity.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Frich, MD, PhD, Principal Investigator — University of Oslo; Ole Jacob Nilsen, MD, Principal Investigator — University of Oslo; Thomas Glott, MD, Principal Investigator — Sunnaas Rehabilitation Hospital, Norway
Locations (2):
- Norway (2):
  - Sunnaas Hospital, Nesoddtangen
  - Oslo University Hospital, Oslo